CLINICAL TRIAL: NCT03303638
Title: Investigating the Impact of Multi-sensory Environments on Behavior During Assisted Bathing for Veterans With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201700547
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Dementia; BPSD
Keywords: Multi-sensory environment; Snoezelen; Bathing; Showering; Tub Bathing
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-sensory Environment during bathing (Other): The MSE intervention will be provided by an interactive waterproof fiber optic kit that includes: a light-emitting diode (LED) wall-washer light, a waterproof fiber optic cable that can be controlled by a waterproof switch held by the participant while bathing, showering, and or tub bathing, and a mobile MSE cart. The wall-washer LED light creates the illusion that the room is painted a variety of bright colors that can be changed by the veteran being bathed. The mobile MSE cart includes an LED solar projector providing visual sensory stimulation by projecting scenes on the wall, an aroma therapy diffuser and a portable bubble tube to create positive distraction during the bathing process.
  Interventions: Behavioral: Multi-sensory Environment

INTERVENTIONS:
Behavioral: Multi-sensory Environment — Multi-sensory environments (MSE), also known as Snoezelen® environments, are defined as behavioral environmental intervention to help people with cognitive and physical impairments reach sensory equilibrium. Typical elements within MSE include visual, auditory, tactile and olfactory stimuli, ergonomic vibro-acoustic furniture, bubble tubes, color-changing LED lighting solutions, music, fiber optics and aromatherapy.

SUMMARY:
Behavioral and psychological symptoms of dementia (BPSD) greatly impact quality of life (QoL) for people with dementia, and pharmacological interventions are costly, ineffective or life-threatening. Law-makers support non-pharmacological interventions like multi-sensory environments (MSE) but they have not been widely studied. There is a critical need for investigation of MSE, particularly during assisted bathing, showering, and/or tub bathing, where most BPSD occur.

DETAILED DESCRIPTION:
Dementia is a debilitating and increasingly pervasive condition impacting cognitive decline across the globe. Behavioral and psychological symptoms of dementia (BPSD) impact quality of life (QoL) for people with dementia and are key interventional targets. Pharmacological interventions for BPSD can be costly, ineffective or life-threatening prompting law makers and the Federal Drug Administration (FDA) to support non-pharmacological interventions like multi-sensory environments (MSE) as the preferred first line of treatment. Despite this support for non-pharmacological interventions like MSE, there has been inconsistency in evaluative methodologies and application of MSE interventions, impeding the widespread use of MSE in dementia-care settings. Therefore, there is a critical need for empirical investigation of well-defined MSE in non-pharmacological dementia-care. The purpose of this study is to investigate the impact of MSE on aggression/agitation during assisted bathing, showering and/or tub bathing for veterans with dementia. The VA has implemented MSE therapy for veterans with dementia since 2010 and the impact of MSE on aggression remains to be evaluated. In 2013, due to favorable initial results, the VA installed both fixed-room and mobile cart MSE applications in 53 VA community living centers (CLCs) across the US, including one in Lake City, Florida which received mobile MSE carts and waterproof MSE equipment for use during assisted bathing, showering, and/or tub bathing. Most acts of aggression/agitation for people with dementia occur during assisted bathing and there is a strong need for evidence-based research of non-pharmacological interventions to reduce problem behaviors, decrease healthcare provider burden and improve quality of life (QoL) for people with dementia. The overall goal of this study is to investigate the effectiveness of MSE in the reduction of agitation/aggression during assisted bathing, showering, and/or tub bathing for veterans with dementia.

ELIGIBILITY:
Veterans being bathed and the healthcare providers providing the bath will be consented in this study.

Inclusion Criteria Veteran with dementia: A veteran with dementia is eligible to participate if they meet the following inclusion criteria:

1. Medical diagnosis of advanced stage dementia (MMSE rating 0-20)
2. Residing within the VA CLC in Lake City, Florida for at least three months
3. Consistently demonstrate high levels of aggression/agitation during assisted bathing, showering, and/or tub bathing.
4. Must have legally authorized representative (LAR) on record

Exclusion criteria Veteran with dementia: A veteran with dementia is ineligible to participate if they meet one of the following exclusion criteria:

1. Predominant diagnosis of psychosis including schizophrenia
2. Patients whom care staff believe would not benefit from MSE.

Inclusion Criteria VA healthcare provider: VA healthcare provider is eligible to participate if they meet the following inclusion criteria:

1. Provides assisted bathing, showering, and/or tub bathing to veterans with dementia at the VA CLC in Lake City, Florida
2. Has worked at the VA CLC in Lake City, Florida for at least three months
3. Speaks English

Exclusion criteria VA healthcare provider: VA healthcare provider is ineligible to participate if they meet one of the following exclusion criteria:

1. Has any limitations that will prevent him/her from providing assisted bathing, showering, and/or tub bathing within a MSE
2. Has any condition which could, in the opinion of the investigator, place the participating veteran at risk or interfere with data integrity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Behavior during assisted bathing | 20 weeks
  Physically aggressive behaviors will be weighted per a three-level category scale: actual, attempted or none.

SECONDARY OUTCOMES:
Impact of MSE related to medication use | 20 weeks
  Scatter plots indicating daily medication use will be overlaid with scatter plots indicating behavior to assess impact of MSE related to medication use.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald I Shorr, MD, Principal Investigator — University of Florida & Veterans Health Administration
Locations (2):
- United States (2):
  - Geriatric Research Education and Clinical Center, Gainesville, Florida
  - Lake City VA Medical Center, Lake City, Florida

IPD SHARING:
Plan to Share IPD: No
Per VA regulations, all data will be stored securely or a server behind VA firewall, only accessible to VA researchers assigned to this study. All data will be de-identified and no names will be referenced in any publications.